CLINICAL TRIAL: NCT07020494
Title: A Randomized, Triple-blind, Placebo Controlled, Parallel Clinical Trial Investigating the Efficacy and Safety of a Lipase Thera-blend and a Lipase Thera-blend + Tributyrin on Memory in Healthy Adults With Self-reported Memory Problems
Brief Title: A Clinical Trial Investigating the Efficacy and Safety of a Lipase Thera-blend and a Lipase Thera-blend + Tributyrin on Memory in Healthy Adults With Self-reported Memory Problems
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Enzymedica (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24EMCFA01
Record Dates: First submitted 2025-05-26; First posted 2025-06-13 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-05

CONDITIONS: Self-reported Memory Problems; Memory
Keywords: Memory; Lipase; Enzyme; Therablend; Tributyrin
MeSH Terms: interventions — tributyrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lipase Thera-blend (Experimental): Lipase Thera-blend consists of lipase from Candida rugosa and lipase from Rhizopus oryzae
  Interventions: Dietary Supplement: Lipase Thera-blend
- Lipase Thera-blend + tributyrin (Experimental): Lipase Thera-blend + tributyrin consists of tributyrin and lipase from Candida rugosa and lipase from Rhizopus oryzae.
  Interventions: Dietary Supplement: Lipase Thera-blend + tributyrin
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lipase Thera-blend — Participants will be instructed to consume take one capsule three times a day with food for the duration of the study period.
  Arms: Lipase Thera-blend
Dietary Supplement: Lipase Thera-blend + tributyrin — Participants will be instructed to consume take one capsule three times a day with food for the duration of the study period.
  Arms: Lipase Thera-blend + tributyrin
Other: Placebo — Participants will be instructed to consume take one capsule three times a day with food for the duration of the study period.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to investigate the efficacy and safety of Lipase Thera-blend and Lipase Thera-blend + tributyrin on memory in healthy adults with self-reported memory problems. The main question[s] it aims to answer [is/are]:

Does of Lipase Thera-blend improve memory in healthy adults? Does Lipase Thera-blend + tributyrin improve memory in healthy adults?

Researchers will compare Lipase Thera-blend and Lipase Thera-blend + tributyrin against a placebo to see if the investigational products improve memory parameters.

Participants will be asked to consume either placebo, Lipase Thera-blend, or Lipase Thera-blend + tributyrin and asked to complete memory questionnaires to assess memory.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 30 and 79 years of age inclusive
2. Females not of child-bearing potential, defined as those who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening

   Or,

   Individuals of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle and agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
   * Abstinence and agrees to use contraception if planning on becoming sexually active during the study
3. Individuals with self-reported memory problems as assessed by a combination score of ≥ 6 on Everyday Memory Questionnaire (EMQ) questions 1, 2 and 18 at screening
4. Absence of dementia or other significant cognitive impairment as assessed by Mini Mental State Examination - 2 Standard Version (MMSE-2) score ≥ 24
5. Agrees to avoid high sources of caffeine (e.g., supplements, tea, coffee, energy drinks) and alcohol consumption for 24 hours prior to in-clinic visits
6. Agrees to avoid first generation anti-allergy medication for 48 hours prior to in-clinic visits
7. Willingness to complete questionnaires, records and diaries associated with the study and to complete all clinic visits
8. Agrees to maintain current lifestyle habits (diet, physical activity, medications, supplements, smoking and sleep) as much as possible throughout the study
9. Provided voluntary, written, informed consent to participate in the study
10. Healthy as determined by medical history and laboratory results as assessed by Qualified Investigator (QI)

Exclusion Criteria:

1. Individuals who are pregnant, breast feeding, or planning to become pregnant during the study
2. Allergy, sensitivity, intolerance, or dietary restriction preventing consumption of investigational product or placebo ingredients
3. Self-reported confirmation of any significant neuropsychological condition and/or cognitive impairment (e.g., Schizophrenia, bipolar disorder, post-traumatic stress disorder, brain injury, stroke, neurodegenerative disease, infections, insomnia, depression, epileptic or other seizure-related disorders) that could interfere with study participation as assessed by the QI
4. Self-reported color blindness/weakness as assessed by the QI
5. Unstable metabolic disease or chronic diseases as assessed by the QI
6. Current or history of any significant diseases of the gastrointestinal tract as assessed by the QI
7. Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the QI (See Section 7.3)
8. Type I diabetes
9. Type II diabetes if on insulin treatment. Type II diabetics on stable medication for at least three months and an HbA1c of <8.0% may be included after assessment by the QI on a case-by-case basis
10. Significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case-by-case basis
11. History of or current diagnosis with kidney, pancreatic, and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones in participants who are symptom free for 6 months
12. Self-reported confirmation of current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
13. Major surgery in the past 3 months or individuals who have planned surgery during the course of the study. Participants with minor surgery will be considered on a case-by-case basis by the QI
14. Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
15. Individuals with an autoimmune disease or are immune compromised
16. Self-reported confirmation of a HIV-, Hepatitis B- and/or C-positive diagnosis as assessed by the QI
17. Self-reported confirmation of blood/bleeding disorders as assessed by the QI
18. Use of medical cannabinoid products
19. Chronic use of cannabinoid products (>2 times/week). Occasional users will be required to washout and abstain for the duration of the study period
20. Alcohol intake average of >2 standard drinks per day as assessed by the QI
21. Alcohol or drug abuse within the last 12 months
22. Current use of prescribed and/or over-the-counter (OTC) medications, supplements, and/or consumption of food/drinks that may impact the efficacy and/or safety of the investigational product (Sections 7.3.1 and 7.3.2)
23. Clinically significant abnormal laboratory results at screening as assessed by the QI
24. Blood donation 30 days prior to baseline, during the study, or a planned donation within 30 days of the last study visit
25. Participation in other clinical research studies 30 days prior to baseline, as assessed by the QI
26. Individuals who are unable to give informed consent
27. Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
The difference in change in spatial, working, and episodic/verbal memory | Day 0 to 84
  The difference in change in spatial, working, and episodic/verbal memory as assessed by the Computerized Mental Performance Assessment System (COMPASS) between Lipase Thera-blend, Lipase Thera-blend + tributyrin and placebo from baseline at day 84. Scoring is not conducted on a scale.
The difference in change in change in memory | Day 0 to 84
  The difference in change in memory as measured by the Everyday Memory Questionnaire (EMQ) between Lipase Thera-blend, Lipase Thera-blend + tributyrin and placebo from baseline at day 84. Reporting is on a scale of 0 to 4, with 0 being "never" (good outcome) and 4 being "several times a day" (worse outcome).

SECONDARY OUTCOMES:
The difference in change in cognition, attention and learning | Day 0 to 84
  The difference in change in cognition, attention and learning as assessed by the Computerized Mental Performance Assessment System (COMPASS) between Lipase Thera-blend, Lipase Thera-blend + tributyrin, and placebo from baseline at day 84
The difference in change in gastrointestinal symptoms | Day 0 to 84
  The difference in change in gastrointestinal symptoms, as assessed by Modified Gastrointestinal Symptom Rating Scale (GSRS) between Lipase Thera-blend, Lipase Thera-blend + tributyrin, and placebo from baseline at day 84. Reporting is on a scale of 0 to 3, with 0 being "no" (good outcome) and 3 being "continuous/frequent/daily" (worse outcome).
The difference in product perception | Day 0 to 84
  The difference in product perception, as assessed by the Product Perception Questionnaire (PPQ) between Lipase Thera-blend, Lipase Thera-blend + tributyrin, and placebo at day 84. Product perception is not scored on a scale.

OTHER OUTCOMES:
Incidence of post-emergent adverse events (AE) | Day 0 to 84
  Incidence of post-emergent adverse events (AE)
Clinically relevant changes in blood pressure after supplementation Indicating an adverse event | Day 0 to 84
  Clinically relevant changes in blood pressure after supplementation Indicating an adverse event
Clinically relevant changes in heart rate after supplementation indicating an adverse event | Day 0 to 84
  Clinically relevant changes in heart rate after supplementation indicating an adverse event
Clinically relevant changes in aspartate aminotransferase (AST) after supplementation indicating an adverse event | Day 0 to 84
  Clinically relevant changes in aspartate aminotransferase (AST) after supplementation indicating an adverse event
Clinically relevant changes in alanine aminotransferase (ALT) after supplementation indicating an adverse event | Day 0 to 84
  Clinically relevant changes in alanine aminotransferase (ALT) after supplementation indicating an adverse event
Clinically relevant changes in alkaline phosphatase (ALP) after supplementation indicating an adverse event | Day 0 to 84
  Clinically relevant changes in alkaline phosphatase (ALP) after supplementation indicating an adverse event
Clinically relevant changes in total bilirubin after supplementation indicating an adverse event | Day 0 to 84
  Clinically relevant changes in total bilirubin after supplementation indicating an adverse event
Clinically relevant changes in creatinine after supplementation indicating an adverse event | Day 0 to 84
  Clinically relevant changes in creatinine after supplementation indicating an adverse event
Clinically relevant changes in electrolytes (Na, K, Cl) after supplementation indicating an adverse event | Day 0 to 84
  Clinically relevant changes in electrolytes (Na, K, Cl) after supplementation indicating an adverse event
Clinically relevant changes in estimated glomerular filtration rate (eGFR)) after supplementation indicating an adverse event | Day 0 to 84
  Clinically relevant changes in estimated glomerular filtration rate (eGFR)) after supplementation indicating an adverse event

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada